CLINICAL TRIAL: NCT00930683
Title: A Phase 1 Multicenter, Open-label Study to Evaluate the Safety and Tolerability of Single and Multiple Intravenous Doses of MEDI-546, a Fully Human Monoclonal Antibody Directed Against Subunit 1 of the Type I Interferon Receptor, in Adult Subjects With Scleroderma
Brief Title: A Study to Evaluate Safety and Tolerability of Multiple Doses of MEDI-546 in Adult Subjects With Scleroderma
Acronym: MEDI-546
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MI-CP180
Record Dates: First submitted 2009-06-29; First posted 2009-06-30 (Estimated); Last update posted 2012-05-08 (Estimated); Status verified 2012-05

CONDITIONS: Scleroderma
MeSH Terms: conditions — Scleroderma, Diffuse | interventions — anifrolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (9):
- 1 (Other): MEDI-546
  Interventions: Drug: MEDI-546
- 2 (Other): MEDI-546
  Interventions: Drug: MEDI-546
- 3 (Other): MEDI-546
  Interventions: Drug: MEDI-546
- 4 (Other): MEDI-546
  Interventions: Drug: MEDI-546
- 5 (Other): MEDI-546
  Interventions: Drug: MEDI-546
- 6 (Other): MEDI-546
  Interventions: Drug: MEDI-546
- 7 (Other): MEDI-546
  Interventions: Drug: MEDI-546
- 8 (Other): MEDI-546
  Interventions: Drug: MEDI-546
- 9 (Other): MEDI-546
  Interventions: Drug: MEDI-546

INTERVENTIONS:
Drug: MEDI-546 — 0.1 mg/kg MEDI-546 as a single IV dose
  Arms: 1
Drug: MEDI-546 — 0.3 mg/kg MEDI-546 as a single IV dose
  Arms: 2
Drug: MEDI-546 — 1.0 mg/kg MEDI-546 as a single IV dose
  Arms: 3
Drug: MEDI-546 — 3.0 mg/kg MEDI-546 as a single IV dose
  Arms: 4
Drug: MEDI-546 — 10.0 mg/kg MEDI-546 as a single IV dose
  Arms: 5
Drug: MEDI-546 — 0.3 mg/kg MEDI-546 as a weekly IV dose x 4 doses
  Arms: 6
Drug: MEDI-546 — 1.0 mg/kg MEDI-546 as a weekly IV dose x 4 doses
  Arms: 7
Drug: MEDI-546 — 5.0 mg/kg MEDI-546 as a weekly IV dose x 4 doses
  Arms: 8
Drug: MEDI-546 — 20.0 mg/kg MEDI-546 as a single IV dose
  Arms: 9

SUMMARY:
To evaluate the safety and tolerability of a multiple-dosed drug (MEDI-546) in adults with scleroderma.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the safety and tolerability of single and multiple IV doses of MEDI-546 in adult subjects with scleroderma who have skin thickening in an area suitable for repeat biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects ≥ 18 years of age at the time of the first dose of MEDI-546;
* Written informed consent and HIPAA authorization (applies to covered entities in the US only) obtained from the subject or subject's legal representative;
* Must fulfill the American Rheumatism Association (American College of Rheumatology) preliminary classification criteria for systemic sclerosis;
* Has at least moderate skin thickening (score of at least 2 by modified Rodnan Total Skin Score [mRTSS]) in at least one area suitable for repeat biopsy, such as arms, legs, or trunk;
* Women, unless surgically sterile (including tubal ligation) or at least 2 years post-menopausal, must use an effective method of avoiding pregnancy (including oral, injectable, transdermal, or implanted contraceptives, intrauterine device, diaphragm with spermicide, cervical cap, abstinence, and sterile sexual partner) in addition to the use of condoms (male or female condoms with spermicide) from signing of the informed consent through the end of the study. Cessation of birth control after this point should be discussed with a responsible physician. Men, unless surgically sterile, must likewise practice 2 effective methods of birth control (condom with spermicide or abstinence) and must use such precautions from Study Day 0 through the end of the study;
* Ability to complete the study period, including follow-up period through a maximum of Study Day 105; and
* Willing to forego other forms of experimental treatment during study.

Exclusion Criteria:

* History of allergy or reaction to any component of the MEDI-546 formulation;
* Forced vital capacity (FVC) < 60% predicted, diffusing capacity for carbon monoxide (DLCO) < 40% predicted, pulmonary hypertension requiring treatment with endothelin receptor antagonists or prostacyclin analogues, scleroderma renal crisis within the last year, or medically significant malabsorption;
* Have received the following medications within 28 days before entry:

  * Cyclophosphamide at any dose
  * Systemic cyclosporine at any dose
  * Thalidomide at any dose
  * Hydroxychloroquine > 600 mg/day
  * Mycophenolate mofetil > 3 g/day
  * Methotrexate > 25 mg/week
  * Azathioprine > 3 mg/kg/day;
* Have received leflunomide > 20 mg/day within 6 months before entry;
* Have received fluctuating doses of the following within 28 days before entry:

  * Antimalarials
  * Mycophenolate mofetil
  * Methotrexate
  * Leflunomide
  * Azathioprine;
* Have received prednisone > 20 mg/day or in fluctuating doses within 14 days before entry;
* Have received fluctuating doses of nonsteroidal anti-inflammatory drugs (NSAIDs) within 14 days before entry;
* Treatment with any investigational drug therapy within 28 days before entry into the study, B cell-depleting therapies within 12 months before entry, or biologic therapies within 30 days or 5 half-lives of the biologic agent, whichever is longer, before entry into the study;
* In the investigator's opinion, evidence of clinically significant active infection, including ongoing, chronic infection, within 28 days before entry;
* A history of severe viral infection as judged by the investigators, including severe infections of either cytomegalovirus (CMV) or the herpes family such as disseminated herpes, herpes encephalitis, ophthalmic herpes;
* Herpes zoster infection within 3 months before entry;
* Evidence of infection with hepatitis B or C virus, or human immunodeficiency virus (HIV)-1 or HIV-2, or active infection with hepatitis A, as determined by results of testing at screening;
* Vaccination with live attenuated viruses within 28 days before entry;
* Pregnancy (women, unless surgically sterile or at least 2 years post-menopausal, must have a negative serum pregnancy test within 28 days before receiving MEDI-546 and a negative urine pregnancy test on days of MEDI-546 administration before receiving MEDI-546);
* Breastfeeding or lactating women;
* History of primary immunodeficiency;
* History of alcohol or drug abuse < 1 year prior to entry;
* History of cancer except basal cell carcinoma or in situ carcinoma of the cervix treated with apparent success with curative therapy > 1 year prior to entry;
* History of active tuberculosis (TB) infection or latent TB infection without completion of an appropriate course of treatment;
* Newly positive TB skin test (defined as a reaction ≥ 10 mm in diameter if not on systemic immunosuppressive medication or ≥ 5 mm if on systemic immunosuppressive medication) without concomitant prophylactic therapy;
* Elective surgery planned from the time of signing of the informed consent through end of study;
* At screening blood tests (within 28 days before entry), any of the following:

  * Aspartate aminotransferase (AST) > 2.5 x upper limit of the normal range (ULN), unless due to Myositis
  * Alanine aminotransferase (ALT) > 2.5 x ULN
  * Creatinine > 4.0 mg/dL
  * Creatinine > 4.0 mg/dL
  * Neutrophils < 1,500/mm3
  * Platelet count < 50,000/mm3;
* History of any disease, evidence of any current disease (other than scleroderma), any finding upon physical examination, chest x-ray, or any laboratory abnormality that, in the opinion of the investigator or medical monitor, may compromise the safety of the subject in the study or confound the analysis of the study; or
* Any employee of the research site who is involved with the conduct of the study.
* History of vasculitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2009-09; Primary Completion 2010-05 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
The safety and tolerability of MEDI-546 will be assessed primarily by summarizing treatment-emergent AEs and SAEs. | Study Day 84 for single-dose; Study Day 105 for multi-dose

SECONDARY OUTCOMES:
The secondary endpoints of the study are to assess the PK, IM, and PD of single and multiple IV doses of MEDI-546 in adult subjects with scleroderma. | Study Day 84 for single-dose; Study Day 105 for multi-dose

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Yoo, M.D., Study Director — MedImmune LLC
Locations (11):
- United States (11):
  - Research Site, Los Angeles, California
  - Boston University, Boston, Massachusetts
  - Research Site, Ann Arbor, Michigan
  - Research Site, New Brunswick, New Jersey
  - Research Site, Lake Success, New York
  - Research Site, Toledo, Ohio
  - Metroplex Clinical Research Center, Dallas, Texas
  - Research Site, Houston, Texas
  - University of Utah Medical Center, Salt Lake City, Utah
  - Research Site, Salt Lake City, Utah
  - Research Site, Seattle, Washington

REFERENCES:
- [Derived] Goldberg A, Geppert T, Schiopu E, Frech T, Hsu V, Simms RW, Peng SL, Yao Y, Elgeioushi N, Chang L, Wang B, Yoo S. Dose-escalation of human anti-interferon-alpha receptor monoclonal antibody MEDI-546 in subjects with systemic sclerosis: a phase 1, multicenter, open label study. Arthritis Res Ther. 2014 Feb 24;16(1):R57. doi: 10.1186/ar4492. PMID 24559157